CLINICAL TRIAL: NCT03470142
Title: The Comparison Between Traditional Laparoscopy-assisted Surgery and Total Laparoscopic Surgery With no Incision (Natural Orifice Transluminal Endoscopic Surgery，NOSES) in Radical Resection of Colorectal Cancer
Brief Title: The Comparison Between Traditional Laparoscopy-assisted Surgery and NOSES in Radical Resection of Colorectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dong Yang (Other)
Responsible Party: Sponsor-Investigator, Dong Yang, doctor, Jilin University
Organization: Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130001
Record Dates: First submitted 2018-03-04; First posted 2018-03-19 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Laparoscopy-assisted Surgery; Total Laparoscopic Surgery With no Incision (Natural Orifice Transluminal Endoscopic Surgery, NOSES)
Keywords: laparoscopy-assisted surgery; NOSES
MeSH Terms: interventions — Natural Orifice Endoscopic Surgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional laparoscopy-assisted surgery (Active Comparator): The traditional laparoscopic operation undergo and then a small incision(5cm) is made in the middle of the lower abdominal wall to trim the mesangial membrane and remove the specimen. At last the anastomosis operation undergo by the laparoscopic operation.
  Interventions: Procedure: traditional laparoscopy-assisted surgery
- total laparoscopic surgery with no incision (NOSES) (Experimental): The whole procedures undergo by total laparoscopic surgery with no incision in the abdominal wall. The specimen then will be removed through natural orifice such as anal.
  Interventions: Procedure: total laparoscopic surgery with no incision (natural orifice transluminal endoscopic surgery, NOSES)

INTERVENTIONS:
Procedure: traditional laparoscopy-assisted surgery — All surgical procedures will be performed by the surgery team ,which is leaded by professor Sun Dong-Hui and Wang Quan. The traditional laparoscopic operation undergo and then a small incision(5cm) is made in the middle of the lower abdominal wall to trim the mesangial membrane and remove the specimen. At last the anastomosis operation undergo by the laparoscopic operation.
  Arms: traditional laparoscopy-assisted surgery
Procedure: total laparoscopic surgery with no incision (natural orifice transluminal endoscopic surgery, NOSES) — All surgical procedures will be performed by the surgery team ,which is leaded by professor Sun Dong-Hui and Wang Quan. The whole procedures undergo by total laparoscopic surgery with no incision in the abdominal wall. The specimen then will be removed through natural orifice (anal).
  Arms: total laparoscopic surgery with no incision (NOSES)

SUMMARY:
This study is to compare the short-term and long-term outcomes of traditional laparoscopy-assisted surgery and total laparoscopic surgery with no incision (natural orifice transluminal endoscopic surgery, NOSES) for colorectal cancer and to find a better surgical method for patients.

ELIGIBILITY:
Inclusion Criteria:

1. All cases should be diagnosed as rectal or sigmoid colon cancer by histology or cytology. The tumor is 5-20cm from the pectinate line. The clinical stage is T1-2, N0, M0 for rectal cancer and T1-T3, N0-2, M0 for sigmoid colon cancer.
2. Eastern Cooperative Oncology Group (ECOG) scale 0-2
3. Heart, lung, liver, and kidney function can tolerate operation
4. Patients and their families are able to understand and be willing to participate in this clinical study and to sign informed consent.

Exclusion Criteria:

1. history of colorectal malignant disease
2. recent diagnosis of other malignant tumors (except for papillary carcinoma of the thyroid gland and basal cell carcinoma of the skin)
3. patients with intestinal obstruction, intestinal perforation, bleeding requiring emergency surgery
4. a history of abdominal surgery (which makes it difficult to perform laparoscopic procedures), severe systemic disease such as diabetes, severe chronic lung disease, cirrhosis, other malignant diseases
5. combined colorectal multiple carcinomas
6. poor anal function before operation and incontinence of defecation
7. with a history of serious mental illness
8. pregnant or lactating women
9. The researchers believe that the patients are unsuitable to participate in the researchers with other cases. A patient or family refusal to join

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2020-03-20 (Estimated); Study Completion 2022-03-20 (Estimated)

PRIMARY OUTCOMES:
the incidence of complications | one month after surgery
  All postoperative complications in the perioperative period will be classified by the Clavien-Dindo classification.The classification mainly focuses on the medical perspective, with major emphasis on the risk and invasiveness of the therapy used to correct a complication. From light to heavy, it consists of five grades (Ⅰ to Ⅴ)

SECONDARY OUTCOMES:
the operation time | in the perioperative period
  The descriptive name of unit would be minute (min).
the blood loss during the operation | in the perioperative period
  The descriptive name of unit would be millilitre (ml).
Postoperative recovery of intestinal peristalsis | in the perioperative period
  The descriptive name of unit would be hour (h).
Visual Analogue Scale/Score | in the perioperative period
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms.For example, the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain ( from 0 to 10).
the functional outcome of defecation, if there is incontinence | Three months after operation
  Anal incontinence was evaluated using the Wexner Continence Grading Scale , the score being calculated after the patients' completion of a daily defecatory questionnaire. Range is from 0 (normal continence) to 20 (maximum incontinence with maximum disturbance of lifestyle).
3-year disease-free survival | three years after operation
cases converted to laparotomy | in the perioperative period
  The procedure for cases who underwent laparoscopy-assisted surgery or NOSES can not go successfully, and then it will be converted to laparotomy. The number of all those cases should be recorded.
The mean postoperative hospital stay | in the perioperative period
  The descriptive name of unit would be day (d).

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Hui Sun, Doctor, Study Director — The First Hospital of Jilin University
Locations (1):
- the First Hospital of Jilin University, Ch’ang-ch’un, Jilin, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.